CLINICAL TRIAL: NCT02094365
Title: A Randomised, Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics and Antiviral Activity of Multiple Doses of Orally Administered ALS-008176 Against Respiratory Syncytial Virus Infection in the Virus Challenge Model
Brief Title: A Phase 2a Study to Evaluate ALS-008176 in the Virus Challenge Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-8176-502
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALS-008176 (Experimental): ALS-008176 drug substance for oral suspension
  Interventions: Drug: ALS-008176
- vehicle alone (Placebo Comparator): Vehicle alone
  Interventions: Drug: vehicle

INTERVENTIONS:
Drug: ALS-008176
  Arms: ALS-008176
Drug: vehicle
  Arms: vehicle alone

SUMMARY:
This study is designed to compare the antiviral effect of ALS-008176 compared to a placebo control in the respiratory syncytial virus challenge model.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 years, inclusive.
* In good health with no history of major medical conditions
* A total body weight ≥ 50 kg and a body mass index (BMI) of > 18kg/m2.

Exclusion Criteria:

* Acute or chronic medical illness
* Positive for Human Immunodeficiency Virus, Hepatitis B or C
* Nose or nasopharynx abnormalities
* Abnormal lung function

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in viral load measurements. | Baseline to day 12

CONTACTS AND LOCATIONS:
Overall Officials: Hosnieh Fathi, MD, MSc, Principal Investigator — Retroscreen Virology Ltd.
Locations (1):
- Retroscreen Virology Ltd, London, United Kingdom

REFERENCES:
- [Derived] DeVincenzo JP, McClure MW, Symons JA, Fathi H, Westland C, Chanda S, Lambkin-Williams R, Smith P, Zhang Q, Beigelman L, Blatt LM, Fry J. Activity of Oral ALS-008176 in a Respiratory Syncytial Virus Challenge Study. N Engl J Med. 2015 Nov 19;373(21):2048-58. doi: 10.1056/NEJMoa1413275. PMID 26580997